CLINICAL TRIAL: NCT02595450
Title: A Non Interventional Trial of Tarceva Metastatic Non Small Lung Cancer.
Brief Title: A Non-interventional Trial of Erlotinib (Tarceva) Metastatic Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22190
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Erlotinib: Participants with locally advanced or metastatic non-small cell lung cancer will be treated with erlotinib according to the product label. This non-interventional study will not affect by any means the treatment, medical care or monitoring of the participant, since it reports retrospective data, which already exist in the participants' medical files.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Participants with locally advanced or metastatic non-small cell lung cancer will be treated with erlotinib according to the product label. This non-interventional study will not affect by any means the treatment, medical care or monitoring of the participant, since it reports retrospective data, which already exist in the participants' medical files.
  Other Names: Tarceva

SUMMARY:
This is a non-interventional, open label, single arm, multicenter study to assess the safety and efficacy of erlotinib in participants with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* It is the physician's decision to prescribe erlotinib in participants and to document their treatment
* Participants must be candidates for receiving erlotinib for locally advanced or metastatic non-small cell lung cancer according to the product label

Exclusion Criteria:

* Participants will be excluded if safety concerns occurred
* If the participant was not compliant or if the participant would wish to stop erlotinib therapy

Ages: 35 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced or metastatic NSCLC that are planned to receive erlotinib containing regimen according to label will be included in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bludesch, Austria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was physician's decision to prescribe erlotinib in participants and to document their treatment cycles.
Groups:
- Erlotinib: Participants with locally advanced or metastatic non-small cell lung cancer were treated with erlotinib according to the product label. This non-interventional study did not affect by any means the treatment, medical care or monitoring of the participant, since it reported retrospective data, which already existed in the participants' medical files.
Period: Overall Study
Arm/Group | Erlotinib
Started | 299
Treated | 291
Completed | 218
Not Completed | 81
Not completed — Unspecified (only completed 1 cycle) | 73
Not completed — Enrolled, but not treated | 8

BASELINE CHARACTERISTICS:
Population: Analysis population included participants who received at least 1 documented treatment cycle.
Arm/Group | Erlotinib
Number analyzed (Participants) | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 172

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time
Description: Time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. Progression was defined as at least 20 percent (%) increase in the sum of diameters of target lesions, or unequivocal progression of existing non-target lesions. Kaplan-Meier estimates were used for calculating PFS.
Time Frame: Up to 6 years
Population: Analysis population included participants who received at least 2 documented treatment cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 218
months | 4.87 [4.07 to 5.90]

2. Primary Outcome: Percentage of Participants With Best Overall Response
Description: Percentage of participants with best overall response of complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) were reported. Per RECIST Version 1.1: CR was defined as complete disappearance of all target lesions and non-target disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimeter [mm]). No new lesions. PR was defined as greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. PD was defined as at least 20% increase in the sum of diameters of target lesions, or unequivocal progression of existing non-target lesions. SD was defined as not qualifying for CR, PR, PD.
Time Frame: Up to 6 years
Population: Analysis population included participants who received at least 2 documented treatment cycles. Missing data was not reported.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 218
percentage of participants
  CR | 0.92
  PR | 15.14
  SD | 63.76
  PD | 12.39

3. Secondary Outcome: Overall Survival (OS) Time
Description: Time from the start of study treatment to date of death due to any cause. Kaplan-Meier estimates were used for calculating OS.
Time Frame: Up to 6 years
Population: As per the study design, no follow up data was collected and documentation ended with end of erlotinib therapy. Due to less events, median OS was not reached.
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 218
months | NA [NA to NA] — Data was not evaluable because as per the study design, no follow up data was collected and documentation ended with end of erlotinib therapy. Due to less events, median OS was not reached.

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: Analysis population included participants who received at least 1 documented treatment cycle.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 14/291
Other Adverse Events (participants affected / at risk) | 134/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=291)
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 3
Aphthous ulcer (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 11
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 1
Hyperhidrosis (General disorders) | 1
Hypogeusia (Nervous system disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=291)
Rash (Skin and subcutaneous tissue disorders) | 123
Diarrhoea (Gastrointestinal disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.